CLINICAL TRIAL: NCT04407247
Title: Treatment of Immune Checkpoint Inhibitor-Related Colitis With Infliximab or Vedolizumab: A Randomized Trial
Brief Title: Infliximab or Vedolizumab in Treating Immune Checkpoint Inhibitor-Related Colitis in Patients With Genitourinary Cancer or Melanoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0276; NCI-2019-04986 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0276 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Colitis; Lung Non-Small Cell Carcinoma; Malignant Genitourinary System Neoplasm; Malignant Solid Neoplasm; Melanoma
MeSH Terms: conditions — Colitis; Carcinoma, Non-Small-Cell Lung; Urogenital Neoplasms; Melanoma | interventions — Infliximab; CT-P13; vedolizumab; Immunoglobulin G; Disulfides; LDP-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (infliximab) (Active Comparator): Patients receive infliximab IV over 1 hour once at week 0, 2, 6 for a total of 3 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Infliximab
- Arm II (vedolizumab) (Experimental): Patients receive vedolizumab IV over 1 hour at week 0, 2, 6 for a total of 3 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Vedolizumab

INTERVENTIONS:
Biological: Infliximab — Given IV
  Other Names: Avakine; cA2; Remicade; Remsima
  Arms: Arm I (infliximab)
Biological: Vedolizumab — Given IV
  Other Names: Entyvio; Immunoglobulin G1, anti-(human integrin LPAM-1 (lymphocyte Peyer''s patch adhesion molecule 1)) (human-Mus musculus heavy chain), disulfide with human-Mus musculus kappa-chain, dimer; LDP 02; LDP-02; LDP02; MLN0002; MLN02
  Arms: Arm II (vedolizumab)

SUMMARY:
This phase I/II trial studies the side effects of infliximab and vedolizumab and to see how well they work in treating inflammation of the colon (colitis) caused by immune checkpoint inhibitor therapy in patients with cancer of the genital and urinary organs (genitourinary) or melanoma. Monoclonal antibodies, such as infliximab or vedolizumab, may help to treat immunotherapy induced colitis/diarrhea. This study may help to identify the optimal treatment strategy for immune checkpoint inhibitor-related colitis in patients with genitourinary cancer or melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the efficacy of infliximab and vedolizumab for clinical remission/response of immune-related diarrhea and/or colitis.

II. To assess the safety and tolerability of the treatment for immune-mediated diarrhea and/or colitis.

SECONDARY OBJECTIVES:

I. To assess the efficacy of infliximab and vedolizumab for clinical remission/response of IMC at 4 weeks.

II. To assess the success of corticosteroid tapering. III. To measure the recurrence rate after corticosteroid taper.

EXPLORATORY OBJECTIVES:

I. To assess the efficacy of infliximab and vedolizumab to achieve endoscopic remission of immune-related diarrhea and/or colitis.

II. To assess the efficacy of infliximab and vedolizumab to achieve histological remission of immune-related diarrhea and/or colitis.

III. To assess the time duration to achieve the clinical remission/response. IV. To assess the long term outcome of cancer. V. To assess immunological, molecular and microbiome changes in tissue/blood/stool.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive infliximab intravenously (IV) over 1 hour once at week 0, 2, 6 for a total of 3 doses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive vedolizumab IV over 1 hour once at week 0, 2, 6 for a total of 3 doses in the absence of disease progression or unacceptable toxicity.

Patients are followed up weekly for 1 month and then at 2 and 3 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive any type of immune checkpoint inhibitor (ICI) therapy
* Patients with peak grade >= 2 immune-related diarrhea and/or colitis (according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 within 45 days prior to initiation of study treatment (infliximab/ vedolizumab)
* Patients with ability to understand and willingness to sign informed consent
* Patients with genitourinary cancer or melanoma or non-small cell lung cancer
* No concern for active concomitant GI infection for immune-related diarrhea and/or colitis work up at the time of protocol therapy initiation as confirmed by stool tests or as per the treating physician based on clinical presentation
* Patient who has been cleared for enrollment by Infectious Diseases consultant or treating physician if positive infection workup or screening tests (e.g. lifelong positive T-spot due to BCG inoculation, chronic colonization) prior to initiation of diarrhea/colitis treatment

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients with persistent gastrointestinal infection confirmed with positive testing despite completing 5 days of antibiotics
* Patients are on concurrent immunosuppressive therapies other than what will be given for colitis
* Patients with preexisting activehistory of inflammatory bowel disease and/or radiation enterocolitis with active disease status at the time of study treatment initiation
* Pregnant and breastfeeding women, and
* Women of child-bearing potential who have positive urine or serum pregnancy test or refuse to do pregnancy test unless last menstrual cycle was > 1 year prior to consent and/ or clear documentation states that patient is peri- or post-menopausal or there was recent supporting objective evidence of 'no pregnancy' status (e.g. blood or imaging) within 30 days prior to initiation of study treatment
* Patients who develop concurrent non-GI toxicity at the time of study treatment initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission/response rate of immune-mediated colitis (IMC) | At 2 weeks after initiation of infliximab or vedolizumab with corticosteroid taper
  The difference of the remission rate between standard of care (infliximab + corticosteroid) and the treatment with vedolizumab + corticosteroid will be calculated along with the 95% confidence interval.
Treatment-related adverse events | Within 3 months after initiation of infliximab or vedolizumab
  Will follow standard reporting guidelines for adverse events. Safety data will be summarized by category, severity and frequency.

SECONDARY OUTCOMES:
Clinical remission/response rate of IMC | At 4 weeks after initiation of infliximab or vedolizumab with corticosteroid taper
  Will be estimated and compared between the two treatment arms using chi-square test.
Complete weaning of corticosteroid | Within 4 weeks after infliximab or vedolizumab initiation without rebound of IMC
  Will be estimated and compared between the two treatment arms using chi-square test.
Recurrent immune-related diarrhea/colitis | Within 3 months after corticosteroid taper
  Will be estimated and compared between the two treatment arms using chi-square test.

OTHER OUTCOMES:
Endoscopic remission (Mayo Clinic sub-score 0-1) of immune-related diarrhea/colitis | At 4 and 8 weeks after initiation of infliximab or vedolizumab treatment
  Will be compared between the two treatment arms.
Histological remission (resolution of active inflammation) of immune-related diarrhea/colitis | At 8 weeks after initiation of infliximab or vedolizumab treatment
  Will be compared between the two treatment arms.
Time duration to achieve clinical remission/response | From initiation of infliximab or vedolizumab treatment to clinical remission/response or last follow-up, assessed up to 3 months
  Will be estimated using the method of Kaplan and Meier. Comparisons of the time-to-event endpoint by important subgroups will be made using the log-rank tests.
Overall survival | From the initiation of infliximab or vedolizumab treatment till death or last follow-up, assessed up to 3 months
  Will be estimated using the method of Kaplan and Meier.
Change in levels of cytokines in tissue/blood/stool samples | Baseline up to 3 months after infliximab or vedolizumab treatment
  Will be compared using 2-sample t-test.
Change in frequencies of immune cells in tissue/blood/stool samples | Baseline up to 3 months after infliximab or vedolizumab treatment
  Will be compared using 2-sample t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghong Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org